CLINICAL TRIAL: NCT03363854
Title: A Randomised, Double-blind, Placebo-controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Tralokinumab in Combination With Topical Corticosteroids in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Tralokinumab in Combination With Topical Corticosteroids for Moderate to Severe Atopic Dermatitis - ECZTRA 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0162-1339; 2017-002065-21 (EudraCT Number)
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2021-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the subject nor any of the investigator or LEO staff who are involved in the treatment or clinical evaluation and monitoring of the subjects will be aware of the treatment received. The packaging and labelling of the investigational medicinal products (IMPs) will contain no evidence of their identity.
  Since tralokinumab and placebo are visually distinct and not matched for viscosity, IMP will be handled and administered by a qualified, unblinded health-care professional at the site who will not be involved in the management of trial subjects and who will not perform any of the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tralokinumab(initial)responders-> Tralokinumab(continuation A) (Experimental): Week 0 to 16 (initial period):
  Tralokinumab loading SC injection on Day 0 followed by tralokinumab injection regimen A.
  Week 16 to 32 (continuation period):
  Tralokinumab continuation SC injection regimen A.
  Interventions: Drug: Tralokinumab
- Tralokinumab(initial)responders-> Tralokinumab(continuation B) (Experimental): Week 0 to 16 (initial period):
  Tralokinumab loading SC injection on Day 0 followed by tralokinumab injection regimen A.
  Week 16 to 32 (continuation period):
  Tralokinumab continuation SC injection regimen B.
  Interventions: Drug: Tralokinumab
- Tralokinumab(initial)non-respon-> Tralokinumab(continuation A) (Experimental): Week 0 to 16 (initial period):
  Tralokinumab loading SC injection on Day 0 followed by tralokinumab injection regimen A.
  Week 16 to 32 (continuation period):
  Tralokinumab continuation SC injection regimen A.
  Interventions: Drug: Tralokinumab
- Placebo (initial)non-respon-> Tralokinumab(continuation A) (Experimental): Week 0 to 16 (initial period):
  Placebo loading SC injection on Day 0 followed by placebo injection regimen A.
  Week 16 to 32 (continuation period):
  Tralokinumab continuation SC injection regimen A.
  Interventions: Drug: Tralokinumab; Drug: Placebo
- Placebo(initial)responders-> Placebo(continuation A) (Placebo Comparator): Week 0 to 16 (initial period):
  Placebo loading SC injection on Day 0 followed by placebo injection regimen A.
  Week 16 to 32 (continuation period):
  Placebo continuation SC injection regimen A.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tralokinumab — Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous (SC) administration.
  Arms: Placebo (initial)non-respon-> Tralokinumab(continuation A); Tralokinumab(initial)non-respon-> Tralokinumab(continuation A); Tralokinumab(initial)responders-> Tralokinumab(continuation A); Tralokinumab(initial)responders-> Tralokinumab(continuation B)
Drug: Placebo — Placebo contains the same excipients in the same concentration only lacking tralokinumab.
  Arms: Placebo (initial)non-respon-> Tralokinumab(continuation A); Placebo(initial)responders-> Placebo(continuation A)

SUMMARY:
Primary objective:

To demonstrate that tralokinumab in combination with topical corticosteroids (TCS) is superior to placebo in combination with TCS in treating moderate-to-severe atopic dermatitis (AD).

Secondary objectives:

To evaluate the efficacy of tralokinumab in combination with TCS on severity and extent of AD, itch, and health-related quality of life compared with placebo in combination with TCS.

To assess the safety of tralokinumab in combination with TCS when used to treat moderate-to-severe AD for 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above.
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD.
* History of AD for ≥1 year.
* Subjects who have a recent history of inadequate response to treatment with topical medications.
* AD involvement of ≥10% body surface area at screening and baseline.
* Stable dose of emollient twice daily (or more, as needed) for at least 14 days before randomisation.

Exclusion Criteria:

* Subjects for whom TCS are medically inadvisable e.g., due to important side effects or safety risks in the opinion of the investigator.
* Active dermatologic conditions that may confound the diagnosis of AD.
* Use of tanning beds or phototherapy within 6 weeks prior to randomisation.
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroid within 4 weeks prior to randomisation.
* Treatment with TCS, topical calcineurin inhibitors (TCI), or topical phosphodiesterase 4 (PDE-4) inhibitor within 2 weeks prior to randomisation.
* Receipt of any marketed biological therapy (i.e. immunoglobulin, anti- immunoglobulin E) including dupilumab or investigational biologic agents within 3 months or 5 half-lives, whichever is longer prior to randomisation.
* Active skin infection within 1 week prior to randomisation.
* Clinically significant infection within 4 weeks prior to randomisation.
* A helminth parasitic infection within 6 months prior to the date informed consent is obtained.
* Tuberculosis requiring treatment within the 12 months prior to screening.
* Known primary immunodeficiency disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical expert, Study Director — LEO Pharma
Locations (66):
- United States (21):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Danbury Clinical Research, Danbury, Connecticut
  - International Dermatology Research, Miami, Florida
  - L & C Professional Medical Research, Miami, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Medical Dermatology Specialists, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana Clinical Trials Center, Plainfield, Indiana
  - Study Center, Bangor, Maine
  - Respiratory Medicine Research, Ypsilanti, Michigan
  - Mount Sinai West Dermatoogy, New York, New York
  - Wake Research, Raleigh, North Carolina
  - Dermatologists of Greater Columbus, Bexley, Ohio
  - Oregon Dermatology & Research, Portland, Oregon
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
- Belgium (4):
  - University Hospital Antwerp, Antwerp
  - Universitair ziekenhuis Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - LEO Pharma Investigational Site, Loverval
- Canada (10):
  - Institute for Skin Advancement, Calgary, Alberta
  - Skin Care Centre, Vancouver, British Columbia
  - Maritime Medical Research Centre, Bathurst, New Brunswick
  - Eastern Canada Cutaneous Research, Halifax, Nova Scotia
  - CCA Medical Research, Ajax, Ontario
  - Simcoderm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - DermEdge Research, Mississauga, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - XLR8 Medical Research, Windsor, Ontario
- Germany (8):
  - Interdisciplinary Study Association GmbH, Berlin
  - St. Josef-Hospital, Ruhr-Universitet, Bochum
  - Klinik und Poliklinik für Dermatologie und Allergologie, Bonn
  - Klinikum der Johann Wolfgang Goethe-Universität Klinik, Frankfurt am Main
  - MensingDerma Research GmbH, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätshautklinik Kiel, Kiel
  - Universitätsklinikum Tübingen, Tübingen
- Netherlands (6):
  - Amcademic Medical Center, Amsterdam
  - LEO Pharma Investigational Site, Bergen op Zoom
  - LEO Pharma Investigational Site, Groningen
  - Radboud MC, Nijmegen
  - Erasmus MC, Rotterdam, Rotterdam
  - University Medical Centre Utrecht, Utrecht
- Poland (5):
  - Nzoz Med-Laser, Lublin
  - LEO Pharma Investigational Site, Rzeszów
  - Wojskowy Instytut Medyczny, Warsaw
  - Wromedica s.c., Wroclaw
  - Derm Medica Sp.zo.o., Wroclaw
- Spain (5):
  - Hospital General de Alicante, Alicante
  - Hospital Universitari de Bellvitge, Barcelona
  - Fundación Hospital Alcorcón, Madrid
  - Hospital de Pontevedra, Pontevedra
  - Hospital General de Valencia, Valencia
- United Kingdom (7):
  - Addenbooke's Hospital, Cambridge, Cambridgeshire
  - The Princess Alexandra Hospital, Harlow, Essex
  - East Surrey Hospital, Redhill, Surrey
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Russells Hall Hospital, Dudley, West Midlands
  - The Royal Free Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayo T, Silverberg JI, Armstrong A, Guttman-Yassky E, Blauvelt A, Esdaile B, Kabashima K, Gooderham M, Kircik L, Schneider S, Bennike N, von Eyben R, Martel BC, Ropke MA, Katoh N, Alexis AF. Efficacy and Safety of Tralokinumab Across Racial Subgroups in Adults with Moderate-to-Severe Atopic Dermatitis: Post Hoc Analysis of Phase III Trials. Am J Clin Dermatol. 2025 Oct 21. doi: 10.1007/s40257-025-00985-1. Online ahead of print. PMID 41118053
- [Derived] Wiseman M, Benvenuto M, Stromkjaer L, Paludan-Muller A, Ryttig L, Petersen AS, Wollenberg A. Cost-Per-Responder Analysis for Tralokinumab and Dupilumab in Combination with Topical Corticosteroids in Patients with Moderate-To-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Oct 16. doi: 10.1007/s13555-025-01565-1. Online ahead of print. PMID 41102518
- [Derived] Paller AS, Soong W, Boguniewicz M, Geng B, Thyssen JP, Bennike N, Schneider S, Wollenberg A. Effect of tralokinumab on moderate-to-severe atopic dermatitis in patients with atopic comorbidities. Ann Allergy Asthma Immunol. 2025 Oct;135(4):425-433.e4. doi: 10.1016/j.anai.2025.06.022. Epub 2025 Jun 22. PMID 40555305
- [Derived] Blauvelt A, Gooderham M, Bhatia N, Langley RG, Schneider S, Zoidis J, Kurbasic A, Armstrong A, Silverberg JI. Tralokinumab Efficacy and Safety, with or without Topical Corticosteroids, in North American Adults with Moderate-to-Severe Atopic Dermatitis: A Subanalysis of Phase 3 Trials ECZTRA 1, 2, and 3. Dermatol Ther (Heidelb). 2022 Nov;12(11):2499-2516. doi: 10.1007/s13555-022-00805-y. Epub 2022 Sep 24. PMID 36152216
- [Derived] Silverberg JI, Adam DN, Zirwas M, Kalia S, Gutermuth J, Pinter A, Pink AE, Chiricozzi A, Barbarot S, Mark T, Tindberg AM, Weidinger S. Tralokinumab Plus Topical Corticosteroids as Needed Provides Progressive and Sustained Efficacy in Adults with Moderate-to-Severe Atopic Dermatitis Over a 32-Week Period: An ECZTRA 3 Post Hoc Analysis. Am J Clin Dermatol. 2022 Jul;23(4):547-559. doi: 10.1007/s40257-022-00702-2. Epub 2022 Jul 20. PMID 35857179

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the participant gave informed consent, they went through a 2- to 6-week screening period for washout of previous atopic dermatitis medication and disallowed medication. The participant was assigned treatment at Week 0.
Groups:
- Tralokinumab Q2W+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at Week 0 followed by a dose of 300 mg tralokinumab Q2W from Week 2 to Week 16.
- Placebo+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with placebo every second week and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at Week 0 followed by administration of placebo every second week from Week 2 to Week 16.
- Tralokinumab R/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 or a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Tralokinumab R/Q4W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 or a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab every fourth week (Q4W) and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received alternating doses of 300 mg tralokinumab and placebo Q2W from Week 16 to Week 30.
- Tralokinumab NR/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), without a clinical response at Week 16 (NR: non-responder) i.e. not having Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16, and assigned tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Placebo NR/Tralokinumab Q2W+TCS: Participants treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), without a clinical response at Week 16 (NR: non-responder) i.e. not having Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16, and assigned tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Placebo R/Placebo+TCS: Participants treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and assigned placebo Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants were administered placebo Q2W from Week 16 to Week 30.
- Safety Follow-up: Participants who spent any amount of time in the safety follow-up period, independently of the treatment(s) received before. No treatment was administered to the participants during the safety follow-up period. In selected countries, eligible participants who completed treatment could transfer to an open-label long-term extension trial (conducted under a separate protocol) at any any time during the safety follow-up period.
Period: Initial Treatment Period
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS | Tralokinumab R/Q2W+TCS | Tralokinumab R/Q4W+TCS | Tralokinumab NR/Q2W+TCS | Placebo NR/Tralokinumab Q2W+TCS | Placebo R/Placebo+TCS | Safety Follow-up
Started | 253 | 127 | 0 (This treatment group applies to the continuation treatment period (see below).) | 0 (This treatment group applies to the continuation treatment period (see below).) | 0 (This treatment group applies to the continuation treatment period (see below).) | 0 (This treatment group applies to the continuation treatment period (see below).) | 0 (This treatment group applies to the continuation treatment period (see below).) | 0 (This treatment group applies to the safety follow-up period (see below).)
Completed | 235 | 120 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 18 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Period: Continuation Treatment Period
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS | Tralokinumab R/Q2W+TCS | Tralokinumab R/Q4W+TCS | Tralokinumab NR/Q2W+TCS | Placebo NR/Tralokinumab Q2W+TCS | Placebo R/Placebo+TCS | Safety Follow-up
Started (Between the inital and continuation treatment periods, 2 participants discontinued treatment.) | 0 (This treatment group applies to the initial treatment period (see above).) | 0 (This treatment group applies to the initial treatment period (see above).) | 69 | 69 | 95 | 79 | 41 | 0 (This treatment group applies to the safety follow-up period (see below).)
Completed | 0 | 0 | 68 | 65 | 87 | 72 | 38 | 0
Not Completed | 0 | 0 | 1 | 4 | 8 | 7 | 3 | 0
Period: Safety Follow-up Period
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS | Tralokinumab R/Q2W+TCS | Tralokinumab R/Q4W+TCS | Tralokinumab NR/Q2W+TCS | Placebo NR/Tralokinumab Q2W+TCS | Placebo R/Placebo+TCS | Safety Follow-up
Started | 0 (This treatment group applies to the initial treatment period (see above).) | 0 (This treatment group applies to the initial treatment period (see above).) | 0 (This treatment group applies to the continuation treatment period (see above).) | 0 (This treatment group applies to the continuation treatment period (see above).) | 0 (This treatment group applies to the continuation treatment period (see above).) | 0 (This treatment group applies to the continuation treatment period (see above).) | 0 (This treatment group applies to the continuation treatment period (see above).) | 278
Completed (Of the 278 participants who started safety follow-up, 180 transferred to the extension trial.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 216

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS | Total
Number analyzed (Participants) | 253 | 127 | 380
Age, Categorical [Count of Participants; unit: Participants] — In this trial, there were 2 age groups: 18-64 years (corresponding to 'between 18 and 65 years') and 65-84 years (corresponding to '>=65 years').
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 237 | 119 | 356
    >=65 years | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (15.3) | 37.7 (14.8) | 39.1 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 43 | 171
  Male | 125 | 84 | 209
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 203 | 85 | 288
  Race: Black or African American | 23 | 12 | 35
  Race: Asian | 17 | 24 | 41
  Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Race: Other | 9 | 5 | 14
  Race: Hispanic or Latino | 0 | 0 | 0
  Race: Not Hispanic or Latino | 0 | 0 | 0
  Ethnicity: White | 0 | 0 | 0
  Ethnicity: Black or African American | 0 | 0 | 0
  Ethnicity: Asian | 0 | 0 | 0
  Ethnicity: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Ethnicity: Other | 0 | 0 | 0
  Ethnicity: Hispanic or Latino | 25 | 9 | 34
  Ethnicity: Not Hispanic or Latino | 228 | 118 | 346
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 15 | 4 | 19
  Canada | 34 | 26 | 60
  Germany | 42 | 15 | 57
  Netherlands | 9 | 7 | 16
  Poland | 48 | 19 | 67
  Spain | 12 | 15 | 27
  United Kingdom | 21 | 13 | 34
  United States | 72 | 28 | 100
Age at onset of atopic dermatitis [Median (Inter-Quartile Range); unit: years] — Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  years
    number analyzed (Participants) | 253 | 126 | 379
    (all) | 4.0 [1.0 to 18.0] | 2.0 [1.0 to 12.0] | 4.0 [1.0 to 16.0]
Duration of atopic dermatitis [Mean (Standard Deviation); unit: years] — Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  years
    number analyzed (Participants) | 253 | 126 | 379
    (all) | 28.0 (16.5) | 28.7 (15.0) | 28.2 (16.0)
Body surface area with atopic dermatitis [Mean (Standard Deviation); unit: percentage affected] | 47.6 (23.3) | 49.0 (25.9) | 48.1 (24.2)
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — IGA is used to evaluate the severity of atopic dermatitis. It is a 5-point score ranging from 0 (clear) to 4 (severe).
  Participants
    Clear | 0 | 0 | 0
    Almost clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 136 | 66 | 202
    Severe | 116 | 60 | 176
    Missing | 1 | 1 | 2
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: units on a scale] — EASI is used to evaluate the extent and severity of atopic dermatitis. It is a composite score ranging from 0 to 72 with a higher score indicating a more extensive and/or severe condition. Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  units on a scale
    number analyzed (Participants) | 252 | 126 | 378
    (all) | 28.81 (11.97) | 30.42 (12.78) | 29.35 (12.25)
Worst Daily Pruritus numeric rating scale (NRS) (weekly average) [Mean (Standard Deviation); unit: units on a scale] — Worst Daily Pruritus NRS is used by the participant to evaluate their worst itch severity over the past 24 hours. The score ranges from 0 ('no itch') to 10 ('worst itch imaginable'). Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  units on a scale
    number analyzed (Participants) | 251 | 126 | 377
    (all) | 7.67 (1.51) | 7.86 (1.49) | 7.74 (1.51)
Scoring Atopic Dermatitis (SCORAD) [Mean (Standard Deviation); unit: units on a scale] — SCORAD is used to evaluate the extent and severity of atopic dermatitis as well as subjective symptoms. The score ranges from 0 to 103 with a higher score indicating a more extensive and/or severe condition. Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  units on a scale
    number analyzed (Participants) | 252 | 126 | 378
    (all) | 66.95 (13.26) | 68.86 (13.19) | 67.59 (13.25)
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: units on a scale] — DLQI is used by the participant to evaluate the impact of their condition on 10 different aspects of health-related quality of life (HRQoL) over the last week. Each item is scored on a 4-point Likert scale ranging from 0 (not at all/not relevant) to 3 (very much). The total score which is the sum of the 10 items ranges from 0 to 30, with a higher score indicating a poorer HRQoL. Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  units on a scale
    number analyzed (Participants) | 250 | 125 | 375
    (all) | 17.58 (7.07) | 17.19 (7.15) | 17.45 (7.09)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: IGA is used to evaluate the severity of atopic dermatitis. It is a 5-point score ranging from 0 (clear) to 4 (severe).
Time Frame: Week 16
Population: Full analysis set (FAS). Of the 380 participants randomised to initial treatment, 378 were treated. Therefore, the FAS consisted of 378 participants (252 + 126).
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
Participants | 98 | 33
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Participants who achieved IGA 0 or 1 at Week 16 were defined as responders. Participants with missing data at Week 16 or who received rescue medication prior to Week 16 were defined as non-responders, independently of their IGA value at Week 16. The null hypothesis of no difference in response rates between tralokinumab Q2W+TCS and placebo+TCS was tested against the 2-sided alternative that there was a difference; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel — The primary endpoints were tested sequentially at a 5% significance level; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 12.4, 95% CI 2-sided [2.9 to 21.9]

2. Primary Outcome: Participants Achieving at Least 75% Reduction in Eczema Area and Severity Index (EASI) at Week 16
Description: EASI is used to evaluate the extent and severity of atopic dermatitis. It is a composite score ranging from 0 to 72 with a higher score indicating a more extensive and/or severe condition.
Time Frame: Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
Participants | 141 | 45
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Participants who achieved at least 75% reduction in EASI at Week 16 were defined as responders. Participants with missing data at Week 16 or who received rescue medication prior to Week 16 were defined as non-responders, independently of their EASI value at Week 16. The null hypothesis of no difference in response rates between tralokinumab Q2W+TCS and placebo+TCS was tested against the 2-sided alternative that there was a difference; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The primary endpoints were tested sequentially at a 5% significance level; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 20.2, 95% CI 2-sided [9.8 to 30.6]

3. Secondary Outcome: Reduction of Worst Daily Pruritus Numeric Rating Scale (NRS) (Weekly Average) of at Least 4 From Baseline to Week 16
Description: Worst Daily Pruritus NRS is used by the participant to evaluate their worst itch severity over the past 24 hours. The score ranges from 0 ('no itch') to 10 ('worst itch imaginable') on an 11-point scale.
Time Frame: Week 0 to Week 16
Population: Participants in the full analysis set with a Worst Daily Pruritus NRS (weekly average) of at least 4 at baseline (Week 0).
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 249 | 126
Participants | 113 | 43
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Participants meeting the endpoint were defined as responders. Participants with missing data at Week 16 or who received rescue medication prior to Week 16 were defined as non-responders, independently of their Worst daily Pruritus NRS value at Week 16; Test type: Superiority; p = 0.037, Cochran-Mantel-Haenszel — This secondary endpoint was tested after the sequential testing of the primary endpoints, if these showed statistical significance; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 11.3, 95% CI 2-sided [0.9 to 21.6]

4. Secondary Outcome: Change in Scoring Atopic Dermatitis (SCORAD) From Baseline to Week 16
Description: SCORAD is used to evaluate the extent and severity of atopic dermatitis as well as subjective symptoms. The score ranges from 0 to 103 with a higher score indicating a more extensive and/or severe condition.
Time Frame: Week 0 to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
units on a scale | -37.7 (1.25) | -26.8 (1.80)
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included; Test type: Superiority; p < 0.001, Repeated measurements model — This secondary endpoint was tested sequentially using the Holm method for multiplicity adjustment at a 5% significance level after the sequential testing of the primary endpoints and first secondary endpoint, if these showed statistical significance; Difference = -10.9, 95% CI 2-sided [-15.2 to -6.6]

5. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Score From Baseline to Week 16
Description: DLQI is used by the participant to evaluate the impact of their condition on 10 different aspects of health-related quality of life (HRQoL) over the last week. Each item is scored on a 4-point Likert scale ranging from 0 (not at all/not relevant) to 3 (very much). The total score which is the sum of the 10 items ranges from 0 to 30, with a higher score indicating a poorer HRQoL.
Time Frame: Week 0 to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
units on a scale | -11.7 (0.39) | -8.8 (0.56)
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, Repeated measurements model — This secondary endpoint was tested sequentially using the Holm method for multiplicity adjustment at a 5% significance level after sequential testing of the primary endpoints and the first secondary endpoint, if these showed statistical significance; Difference = -2.9, 95% CI 2-sided [-4.3 to -1.6]

6. Secondary Outcome: Frequency of Anti-drug Antibodies (ADA)
Description: Presence of ADA from Week 0 to Week 32 was measured. Data were reported in the following categories: positive (presence of ADA at baseline and/or presence of ADA at at least 1 post-baseline assessment), perishing (presence of ADA at baseline and absence of ADA at all post-baseline assessments), negative (absence of ADA at all assessments), no post-baseline ADA assessment. Perishing ADAs were not assessed in the continuation treatment period.
Time Frame: Week 0 to Week 16, Week 16 to Week 32
Population: Safety analysis set (378 participants). Data was collected for the treatment groups applicable in each treatment period, i.e. tralokinumab Q2W+TCS and placebo+TCS treatment groups in the initial treatment period and the 5 continuation treatment groups (see table below) in the continuation treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Initial Treatment Period - Tralokinumab Q2W+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at Week 0 followed by a dose of 300 mg tralokinumab Q2W from Week 2 to Week 16.
- Initial Treatment Period - Placebo+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with placebo every second week and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at Week 0 followed by administration of placebo every second week from Week 2 to Week 16.
- Continuation Treatment Period - Tralokinumab R/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 or a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Continuation Treatment Period - Tralokinumab R/Q4W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 or a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab every fourth week (Q4W) and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received alternating doses of 300 mg tralokinumab and placebo Q2W from Week 16 to Week 30.
- Continuation Treatment Period - Tralokinumab NR/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), without a clinical response at Week 16 (NR: non-responder) i.e. not having Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16, and assigned tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Continuation Treatment Period - Placebo NR/Tralokinumab Q2W+TCS: Participants treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), without a clinical response at Week 16 (NR: non-responder) i.e. not having Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16, and assigned tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Continuation Treatment Period - Placebo R/Placebo+TCS: Participants treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and assigned placebo Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants were administered placebo Q2W from Week 16 to Week 30.
Arm/Group | Initial Treatment Period - Tralokinumab Q2W+TCS | Initial Treatment Period - Placebo+TCS | Continuation Treatment Period - Tralokinumab R/Q2W+TCS | Continuation Treatment Period - Tralokinumab R/Q4W+TCS | Continuation Treatment Period - Tralokinumab NR/Q2W+TCS | Continuation Treatment Period - Placebo NR/Tralokinumab Q2W+TCS | Continuation Treatment Period - Placebo R/Placebo+TCS
Number analyzed (Participants) | 252 | 126 | 69 | 69 | 95 | 79 | 41
Participants
  Initial treatment period (Week 0 to Week 16): number analyzed (Participants) | 252 | 126 | 0 | 0 | 0 | 0 | 0
  Initial treatment period (Week 0 to Week 16): Positive | 2 | 3 | 0 | 0 | 0 | 0 | 0
  Initial treatment period (Week 0 to Week 16): Perishing | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Initial treatment period (Week 0 to Week 16): Negative | 246 | 123 | 0 | 0 | 0 | 0 | 0
  Initial treatment period (Week 0 to Week 16): No post-baseline ADA assessment | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Continuation treatment period (Week 16 to Week 32): number analyzed (Participants) | 0 | 0 | 66 | 65 | 92 | 77 | 39
  Continuation treatment period (Week 16 to Week 32): Positive | 0 | 0 | 0 | 2 | 0 | 3 | 2
  Continuation treatment period (Week 16 to Week 32): Perishing | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Continuation treatment period (Week 16 to Week 32): Negative | 0 | 0 | 66 | 63 | 92 | 74 | 37
  Continuation treatment period (Week 16 to Week 32): No post-baseline ADA assessment | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Amount of Topical Corticosteroid (TCS) Used Through Week 16 Assuming no TCS Used From the Non-returned Tubes
Description: Assessed as the amount of TCS weighed from previous visits, assuming no TCS was used from the non-returned tubes. Measurements were collected as TCS weight (g) between the visits.
Time Frame: Week 1-2 to Week 15-16
Population: Full analysis set. Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included.
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
g
  Week 1-2: number analyzed (Participants) | 250 | 125
  Week 1-2 | 29.3 (2.45) | 32.8 (3.47)
  Week 3-4: number analyzed (Participants) | 248 | 121
  Week 3-4 | 19.7 (1.86) | 26.6 (2.66)
  Week 5-6: number analyzed (Participants) | 245 | 118
  Week 5-6 | 18.5 (1.72) | 23.2 (2.46)
  Week 7-8: number analyzed (Participants) | 240 | 114
  Week 7-8 | 17.0 (2.04) | 24.3 (2.93)
  Week 9-10: number analyzed (Participants) | 236 | 113
  Week 9-10 | 14.8 (1.66) | 23.9 (2.38)
  Week 11-12: number analyzed (Participants) | 234 | 110
  Week 11-12 | 11.6 (1.38) | 19.6 (2.00)
  Week 13-14: number analyzed (Participants) | 232 | 108
  Week 13-14 | 12.7 (1.61) | 23.0 (2.33)
  Week 15-16: number analyzed (Participants) | 229 | 108
  Week 15-16 | 11.6 (1.57) | 20.2 (2.27)
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 1-2 are reported below; Test type: Superiority; p = 0.41, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -3.5, 95% CI 2-sided [-11.9 to 4.9]
Statistical Analysis 2: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 3-4 are reported below; Test type: Superiority; p = 0.033, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -6.9, 95% CI 2-sided [-13.3 to -0.6]
Statistical Analysis 3: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 5-6 are reported below; Test type: Superiority; p = 0.12, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -4.7, 95% CI 2-sided [-10.6 to 1.2]
Statistical Analysis 4: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 7-8 are reported below; Test type: Superiority; p = 0.043, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -7.3, 95% CI 2-sided [-14.3 to -0.2]
Statistical Analysis 5: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 9-10 are reported below; Test type: Superiority; p = 0.002, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -9.1, 95% CI 2-sided [-14.8 to -3.4]
Statistical Analysis 6: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 11-12 are reported below; Test type: Superiority; p = 0.001, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -8.0, 95% CI 2-sided [-12.8 to -3.2]
Statistical Analysis 7: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 13-14 are reported below; Test type: Superiority; p < 0.001, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -10.2, 95% CI 2-sided [-15.8 to -4.7]
Statistical Analysis 8: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 15-16 are reported below; Test type: Superiority; p = 0.002, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -8.6, 95% CI 2-sided [-14.1 to -3.2]

8. Secondary Outcome: Amount of Topical Corticosteroid (TCS) Used Through Week 16 Assuming All TCS Used From the Non-returned Tubes
Description: Assessed as the amount of TCS weighed from previous visits, assuming all TCS was used from the non-returned tubes. Measurements were collected as TCS weight (g) between the visits.
Time Frame: Week 1-2 to Week 15-16
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
g
  Week 1-2: number analyzed (Participants) | 250 | 125
  Week 1-2 | 40.1 (3.22) | 40.1 (4.57)
  Week 3-4: number analyzed (Participants) | 248 | 121
  Week 3-4 | 32.4 (3.00) | 31.3 (4.27)
  Week 5-6: number analyzed (Participants) | 245 | 118
  Week 5-6 | 29.2 (2.89) | 30.6 (4.13)
  Week 7-8: number analyzed (Participants) | 240 | 114
  Week 7-8 | 25.2 (2.89) | 30.0 (4.15)
  Week 9-10: number analyzed (Participants) | 236 | 113
  Week 9-10 | 22.5 (2.61) | 26.9 (3.76)
  Week 11-12: number analyzed (Participants) | 234 | 110
  Week 11-12 | 16.9 (2.23) | 23.1 (3.22)
  Week 13-14: number analyzed (Participants) | 232 | 108
  Week 13-14 | 16.6 (2.22) | 25.5 (3.23)
  Week 15-16: number analyzed (Participants) | 229 | 108
  Week 15-16 | 15.3 (2.26) | 24.8 (3.27)
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 1.00, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.0, 95% CI 2-sided [-11.0 to 11.0]
Statistical Analysis 2: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.83, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 1.1, 95% CI 2-sided [-9.1 to 11.4]
Statistical Analysis 3: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.78, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -1.4, 95% CI 2-sided [-11.3 to 8.5]
Statistical Analysis 4: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.34, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -4.8, 95% CI 2-sided [-14.8 to 5.1]
Statistical Analysis 5: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 5]; Test type: Superiority; p = 0.34, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -4.4, 95% CI 2-sided [-13.4 to 4.6]
Statistical Analysis 6: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 6]; Test type: Superiority; p = 0.11, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -6.2, 95% CI 2-sided [-13.9 to 1.5]
Statistical Analysis 7: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 7]; Test type: Superiority; p = 0.024, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -8.9, 95% CI 2-sided [-16.6 to -1.2]
Statistical Analysis 8: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 7, analysis 8]; Test type: Superiority; p = 0.017, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -9.5, 95% CI 2-sided [-17.3 to -1.7]

9. Secondary Outcome: Number of Atopic Dermatitis Flares Through Week 16
Description: Assessed as appearance of new flares since previous visit.
Time Frame: Week 0 to Week 16
Population: Full analysis set. All observed data
Measure: Number; unit: number of flares
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
number of flares | 119 | 75

10. Secondary Outcome: Number of Days Without Topical Treatment Use From Baseline to Week 16
Description: Participants assessed their use of topical treatment over the past 24 hours using a response scale ('yes', 'no'). Measurements of number of days per week were used in the analysis.
Time Frame: Week 1 to Week 16
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
days
  Week 1: number analyzed (Participants) | 210 | 99
  Week 1 | 2.6 (0.17) | 2.5 (0.25)
  Week 2: number analyzed (Participants) | 208 | 98
  Week 2 | 3.0 (0.18) | 2.6 (0.27)
  Week 3: number analyzed (Participants) | 219 | 104
  Week 3 | 2.9 (0.17) | 2.7 (0.25)
  Week 4: number analyzed (Participants) | 220 | 98
  Week 4 | 3.1 (0.17) | 2.7 (0.25)
  Week 5: number analyzed (Participants) | 217 | 97
  Week 5 | 3.2 (0.17) | 2.7 (0.25)
  Week 6: number analyzed (Participants) | 216 | 102
  Week 6 | 3.1 (0.18) | 2.8 (0.26)
  Week 7: number analyzed (Participants) | 209 | 96
  Week 7 | 3.3 (0.17) | 2.7 (0.25)
  Week 8: number analyzed (Participants) | 208 | 97
  Week 8 | 3.3 (0.18) | 3.0 (0.26)
  Week 9: number analyzed (Participants) | 217 | 98
  Week 9 | 3.6 (0.17) | 2.6 (0.25)
  Week 10: number analyzed (Participants) | 217 | 96
  Week 10 | 3.4 (0.17) | 2.7 (0.25)
  Week 11: number analyzed (Participants) | 213 | 97
  Week 11 | 3.6 (0.18) | 2.7 (0.26)
  Week 12: number analyzed (Participants) | 218 | 97
  Week 12 | 3.4 (0.18) | 2.7 (0.26)
  Week 13: number analyzed (Participants) | 216 | 95
  Week 13 | 3.5 (0.18) | 2.7 (0.26)
  Week 14: number analyzed (Participants) | 206 | 98
  Week 14 | 3.3 (0.18) | 2.6 (0.26)
  Week 15: number analyzed (Participants) | 207 | 97
  Week 15 | 3.5 (0.18) | 2.8 (0.26)
  Week 16: number analyzed (Participants) | 210 | 96
  Week 16 | 3.4 (0.19) | 3.0 (0.27)
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 1 are reported below; Test type: Superiority; p = 0.64, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 2: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 2 are reported below; Test type: Superiority; p = 0.26, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.4, 95% CI 2-sided [-0.3 to 1.0]
Statistical Analysis 3: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 3 are reported below; Test type: Superiority; p = 0.46, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.2, 95% CI 2-sided [-0.4 to 0.8]
Statistical Analysis 4: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 4 are reported below; Test type: Superiority; p = 0.16, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.4, 95% CI 2-sided [-0.2 to 1.0]
Statistical Analysis 5: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 5 are reported below; Test type: Superiority; p = 0.13, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.5, 95% CI 2-sided [-0.1 to 1.1]
Statistical Analysis 6: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 6 are reported below; Test type: Superiority; p = 0.38, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.3, 95% CI 2-sided [-0.3 to 0.9]
Statistical Analysis 7: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 7 are reported below; Test type: Superiority; p = 0.040, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.6, 95% CI 2-sided [0.0 to 1.2]
Statistical Analysis 8: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 8 are reported below; Test type: Superiority; p = 0.31, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.3, 95% CI 2-sided [-0.3 to 1.0]
Statistical Analysis 9: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 9 are reported below; Test type: Superiority; p = 0.001, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 1.0, 95% CI 2-sided [0.4 to 1.6]
Statistical Analysis 10: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 10 are reported below; Test type: Superiority; p = 0.026, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.7, 95% CI 2-sided [0.1 to 1.3]
Statistical Analysis 11: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 11 are reported below; Test type: Superiority; p = 0.006, Repeated measurements model] — The statistical test was not controlled for multiplicity; Difference = 0.9, 95% CI 2-sided [0.2 to 1.5]
Statistical Analysis 12: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 12 are reported below; Test type: Superiority; p = 0.043, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.6, 95% CI 2-sided [0.0 to 1.3]
Statistical Analysis 13: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 13 are reported below; Test type: Superiority; p = 0.010, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.8, 95% CI 2-sided [0.2 to 1.4]
Statistical Analysis 14: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 14 are reported below; Test type: Superiority; p = 0.037, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.7, 95% CI 2-sided [0.0 to 1.3]
Statistical Analysis 15: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 15 are reported below; Test type: Superiority; p = 0.045, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.6, 95% CI 2-sided [0.0 to 1.3]
Statistical Analysis 16: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Data collected after permanent discontinuation of investigational medicinal product or initiation of rescue medication were not included. Results of Week 16 are reported below; Test type: Superiority; p = 0.17, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = 0.5, 95% CI 2-sided [-0.2 to 1.1]

11. Secondary Outcome: Participants Achieving at Least 50% Reduction in Eczema Area and Severity Index (EASI) at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
Participants | 200 | 73
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Participants meeting the endpoint were defined as responders. Participants with missing data at Week 16 or who received rescue medication prior to Week 16 were defined as non-responders, independently of their EASI value at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The statistical test was not controlled for multiplicity; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 21.3, 95% CI 2-sided [11.3 to 31.3]

12. Secondary Outcome: Participants Achieving at Least 90% Reduction in Eczema Area and Severity Index (EASI) at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
Participants | 83 | 27
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel — The statistical test was not controlled for multiplicity; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 11.4, 95% CI 2-sided [2.1 to 20.7]

13. Secondary Outcome: Change From Baseline to Week 16 in Eczema Area and Severity Index (EASI) Score
Description: as for outcome 2
Time Frame: Week 0 to Week 16
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 229 | 108
units on a scale | -21.0 (0.67) | -15.6 (0.96)
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, Repeated measurement model — The statistical test was not controlled for multiplicity; Difference = -5.4, 95% CI 2-sided [-7.7 to -3.1]

14. Secondary Outcome: Participants Achieving at Least 50% Reduction in Scoring Atopic Dermatitis (SCORAD) at Week 16
Description: as for outcome 4
Time Frame: Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
Participants | 154 | 48
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Partcipants meeting the endpoint were defined as responders. Participants with missing data at Week 16 or who received rescue medication prior to Week 16 were defined as non-responders, independently of their SCORAD value at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The statistical test was not controlled for multiplicity; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 22.9, 95% CI 2-sided [12.4 to 33.3]

15. Secondary Outcome: Participants Achieving at Least 75% Reduction in Scoring Atopic Dermatitis (SCORAD) at Week 16
Description: as for outcome 4
Time Frame: Week 16
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 252 | 126
Participants | 60 | 16
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Participants meeting the endpoint were defined as responders. Participants with missing data at Week 16 or who received rescue medication prior to Week 16 were defined as non-responders, independently of their SCORAD value at Week 16; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel — The statistical test was not controlled for multiplicity; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 11.1, 95% CI 2-sided [3.2 to 19.0]

16. Secondary Outcome: Change From Baseline to Week 16 in Worst Daily Pruritus Numeric Rating Scale (NRS) (Weekly Average)
Description: as for outcome 3
Time Frame: Week 0 to Week 16
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 221 | 100
units on a scale | -4.1 (0.15) | -2.9 (0.21)
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, Repeated measurements model — The statistical test was not controlled for multiplicity; Difference = -1.2, 95% CI 2-sided [-1.7 to -0.7]

17. Secondary Outcome: Reduction From Baseline to Week 16 of Dermatology Life Quality Index (DLQI) of at Least 4 Points Among Participants With Baseline DLQI ≥4
Description: as for outcome 5
Time Frame: Week 0 to Week 16
Population: Participants in the full analysis set with DLQI of at least 4 at baseline (Week 0).
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab Q2W+TCS | Placebo+TCS
Number analyzed (Participants) | 248 | 123
Participants | 207 | 81
Statistical Analysis 1: Comparison: Tralokinumab Q2W+TCS vs Placebo+TCS; Participants meeting the endpoint were defined as responders. Participants with missing data at Week 16 or who received rescue medication prior to Week 16 were defined as non-responders, independently of their DLQI value at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The statistical test was not controlled for multiplicity; The analysis was conducted using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Risk Difference (RD) = 17.6, 95% CI 2-sided [8.0 to 27.1]

18. Secondary Outcome: Participants With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 32 Among Participants With IGA Score of 0 or 1 at Week 16 After Initial Randomisation to Tralokinumab
Description: IGA is used to evaluate the severity of atopic dermatitis. It is a 5-point score ranging from 0 (clear) to 4 (severe).
Time Frame: Week 32
Population: Participants in the continuation treatment analysis set treated with tralokinumab Q2W+TCS in the initial treatment period and who achieved IGA score of 0 or 1 at Week 16 without rescue medication. Participants who received rescue medication prior to Week 32 or with missing data at Week 32 were not included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Tralokinumab R/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as IGA score of 0 or 1 at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Tralokinumab R/Q4W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as IGA score of 0 or 1 at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab every fourth week (Q4W) and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received alternating doses of 300 mg tralokinumab and placebo Q2W from Week 16 to Week 30.
Arm/Group | Tralokinumab R/Q2W+TCS | Tralokinumab R/Q4W+TCS
Number analyzed (Participants) | 48 | 49
Participants | 43 | 38

19. Secondary Outcome: Participants Achieving at Least 75% Reduction in Eczema Area and Severity Index (EASI) at Week 32 Among Participants Who Had Achieved at Least 75% Reduction in EASI at Week 16 After Initial Randomisation to Tralokinumab
Description: as for outcome 2
Time Frame: Week 32
Population: Participants in the continuation treatment analysis set treated with tralokinumab Q2W+TCS in the initial treatment period and who achieved at least 75% reduction in EASI at Week 16 without rescue medication. Participants who received rescue medication prior to Week 32 or with missing data at Week 32 were not included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Tralokinumab R/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as a reduction in EASI of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Tralokinumab R/Q4W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as a reduction in EASI of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab every fourth week (Q4W) and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received alternating doses of 300 mg tralokinumab and placebo Q2W from Week 16 to Week 30.
Arm/Group | Tralokinumab R/Q2W+TCS | Tralokinumab R/Q4W+TCS
Number analyzed (Participants) | 67 | 65
Participants | 62 | 59

ADVERSE EVENTS:
Time Frame: Initial treatment period (Week 0 to Week 16), continuation treatment period (Week 16 to Week 32), safety follow-up (Week 32 to Week 46).
Description: The analysis was conducted based on the safety analysis set which consisted of subjects exposed to at least 1 dose of investigational medicinal product.
Groups:
- Initial Treatment Period: Tralokinumab Q2W+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at Week 0 followed by a dose of 300 mg tralokinumab Q2W from Week 2 to Week 16.
- Initial Treatment Period: Placebo+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with placebo every second week and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at Week 0 followed by administration of placebo every second week from Week 2 to Week 16.
- Continuation Treatment Period: Tralokinumab R/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 or a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Continuation Treatment Period: Tralokinumab R/Q4W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 or a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and re-randomised to tralokinumab every fourth week (Q4W) and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received alternating doses of 300 mg tralokinumab and placebo Q2W from Week 16 to Week 30.
- Continuation Treatment Period: Tralokinumab NR/Q2W+TCS: Participants treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), without a clinical response at Week 16 (NR: non-responder) i.e. not having Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16, and assigned tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Continuation Treatment Period: Placebo NR/Tralokinumab Q2W+TCS: Participants treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), without a clinical response at Week 16 (NR: non-responder) i.e. not having Investigator's Global Assessment score of 0 or 1 at Week 16 nor a reduction in Eczema Area and Severity Index of at least 75% at Week 16, and assigned tralokinumab Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants received a dose of 300 mg tralokinumab Q2W from Week 16 to Week 30.
- Continuation Treatment Period: Placebo R/Placebo+TCS: Participants treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed in the initial treatment period (Week 0 to Week 16), with a clinical response at Week 16 (R: responder) defined as Investigator's Global Assessment score of 0 or 1 at Week 16 or a reduction in Eczema Area and Severity Index of at least 75% at Week 16 achieved without rescue treatment, and assigned placebo Q2W and TCS as needed in the continuation treatment period (Week 16 to Week 32).
  Participants were administered placebo Q2W from Week 16 to Week 30.
Arm/Group | Initial Treatment Period: Tralokinumab Q2W+TCS | Initial Treatment Period: Placebo+TCS | Continuation Treatment Period: Tralokinumab R/Q2W+TCS | Continuation Treatment Period: Tralokinumab R/Q4W+TCS | Continuation Treatment Period: Tralokinumab NR/Q2W+TCS | Continuation Treatment Period: Placebo NR/Tralokinumab Q2W+TCS | Continuation Treatment Period: Placebo R/Placebo+TCS | Safety Follow-up
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/126 | 0/69 | 0/69 | 0/95 | 0/79 | 0/41 | 0/278
Serious Adverse Events (participants affected / at risk) | 2/252 | 4/126 | 3/69 | 0/69 | 2/95 | 0/79 | 1/41 | 3/278
Other Adverse Events (participants affected / at risk) | 118/252 | 36/126 | 30/69 | 24/69 | 41/95 | 32/79 | 12/41 | 10/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Treatment Period: Tralokinumab Q2W+TCS (N=252) | Initial Treatment Period: Placebo+TCS (N=126) | Continuation Treatment Period: Tralokinumab R/Q2W+TCS (N=69) | Continuation Treatment Period: Tralokinumab R/Q4W+TCS (N=69) | Continuation Treatment Period: Tralokinumab NR/Q2W+TCS (N=95) | Continuation Treatment Period: Placebo NR/Tralokinumab Q2W+TCS (N=79) | Continuation Treatment Period: Placebo R/Placebo+TCS (N=41) | Safety Follow-up (N=278)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Treatment Period: Tralokinumab Q2W+TCS (N=252) | Initial Treatment Period: Placebo+TCS (N=126) | Continuation Treatment Period: Tralokinumab R/Q2W+TCS (N=69) | Continuation Treatment Period: Tralokinumab R/Q4W+TCS (N=69) | Continuation Treatment Period: Tralokinumab NR/Q2W+TCS (N=95) | Continuation Treatment Period: Placebo NR/Tralokinumab Q2W+TCS (N=79) | Continuation Treatment Period: Placebo R/Placebo+TCS (N=41) | Safety Follow-up (N=278)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 2 (2) | 4 (4) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 17 (30) | 0 (0) | 5 (14) | 4 (9) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 28 (32) | 4 (4) | 4 (4) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 4 (6) | 1 (2) | 3 (3) | 4 (4) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 19 (21) | 6 (7) | 7 (8) | 3 (3) | 6 (7) | 3 (3) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 49 (64) | 14 (18) | 12 (13) | 9 (10) | 20 (28) | 15 (15) | 7 (8) | 0 (0)
Headache (Nervous system disorders) | 22 (26) | 6 (9) | 2 (2) | 5 (5) | 7 (7) | 2 (2) | 1 (1) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (8) | 10 (12) | 1 (1) | 1 (1) | 8 (8) | 6 (7) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all phase 3 clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03363854/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03363854/SAP_001.pdf